CLINICAL TRIAL: NCT02539459
Title: A Phase II Study of Sporadic Angiomyolipomas (AMLs) Growth Kinetics While on Everolimus Therapy
Brief Title: Sporadic Angiomyolipomas (AMLs) Growth Kinetics While on Everolimus
Acronym: SAGE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Extreme toxicity, met toxicity stopping rules
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-070
Record Dates: First submitted 2015-08-20; First posted 2015-09-03 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Sporadic Angiomyolipomas (AMLs)
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (everolimus) (Experimental): Patients will take 10 mg (1 tablet) of everolimus each day for 4 months
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — 10 mg tablets

SUMMARY:
The purpose of this research study is to see if oral everolimus is tolerable and effective in the treatment of sporadic Angiomyolipomas (AMLs). AMLs are the most common non-cancerous tumor of the kidney. They are composed of blood vessels, muscle cells and fat cells.Everolimus is already an approved drug for several other diseases like kidney cancer, but is being studied now specifically to see if it is helpful for people with AML.

DETAILED DESCRIPTION:
Primary Objective

1. To evaluate the efficacy and tolerability of everolimus in reducing tumor volume in sporadic AMLs as measured by dynamic contrast enhanced magnetic resonance imaging (DCE MRI), in patients who might otherwise be considered for active surgical or percutaneous intervention.

Secondary Objectives

1. To evaluate health-related quality of life (HRQoL) in subjects treated with everolimus for sporadic AMLs.
2. To assess the growth kinetics of sporadic AMLs in patients who have been treated with everolimus as part of the study and demonstrate an objective response as well as those who have been treated with everolimus during the study with a suboptimal or no response.
3. To measure the rate of surgical or percutaneous (embolization) intervention at 1 year from day 1 of study.
4. To assess the safety and tolerability of everolimus in patients with sporadic AML.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of renal AML > 3 cm confirmed on pre-enrollment Dynamic Contrast Enhanced MRI (DCE-MRI)
* Must not have received any prior treatment for AML
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Absolute neutrophil count >= 1,500/ microliter (mcL)
* Hemoglobin >=10 g/dL
* Platelets >= 100,000/ mcL
* international normalized ratio (INR) <= 1.2 X Upper limit Normal (ULN)
* activated partial thromboplastin time (aPTT) <= 1.2 X ULN
* aspartate aminotransferase (AST) / alanine transaminase (ALT) <= 2.5 X ULN
* Total bilirubin <= 2.0mg/dL
* Renal Function epidermal growth factor receptor (eGFR) >= 30 mL/min via calculated creatinine clearance
* Fasting serum cholesterol <= 300 mg/dL OR <= 7.75 mmol/L AND fasting triglycerides <= 2.5x ULN.

Exclusion Criteria:

* History of tuberous sclerosis, LAM or any active malignancy
* Treatment with any other investigational agents for any other disease
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding or affect absorption of investigational product
* Active diarrhea of any grade.
* History of human immunodeficiency virus (HIV) infection, hepatitis B or C (screening for all three is mandatory prior to study); prior hepatitis C infection
* Presence of any active or ongoing infection.
* Any known uncontrolled underlying pulmonary disease by history, physical exam or if applicable pulmonary function test (PFTs)
* History of certain cardiovascular conditions within the past 6 months
* History of Class III or IV congestive heart failure, as defined by the New York Heart Association Classification of Congestive Heart Failure.
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Corrected QT interval (QTc) > 480 milliseconds
* Poorly controlled hypertension, defined as systolic blood pressure (SBP) of >= 140 millimeters of mercury(mmHg) or diastolic blood pressure (DBP) of >= 90 mmHg.
* Evidence of active bleeding or bleeding diathesis
* Uncontrolled diabetes mellitus (defined by a Hgb A1c >8) obtained within 14 days prior to registration. Optimal glucose control (Hgb A1c <= 8) must be achieved before registration and monitored during protocol treatment
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications
* Concurrent therapy given to treat cancer including treatment with an investigational agent or concurrent participation in another clinical trial involving anti-cancer investigational drug.
* Administration of any investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to everolimus
* Prior or current use of systemic anti-vascular endothelial growth factor (VEGF) inhibitors, cytokines or mechanistic target of rapamycin (mTOR) inhibitors (e.g. interferon, interleukin 2).
* Pregnant or nursing (lactating) women
* Women of child-bearing potential (WOCBP) must use highly effective methods of contraception during the study and 8 weeks after.
* Unable to obtain a contrast (gadolinium) based DCE MRI, including include patients with pacemakers, automatic implantable cardioverter/defibrillator (AICDs), non MRI compatible metallic implants or eGFR <30.
* Must not have received immunization with an attenuated live vaccine within seven days prior to registration nor have plans to receive such vaccination while on protocol treatment
* Must not be taking, nor plan to take while on protocol treatment, strong cytochrome P450 3A4 (CYP3A4) inhibitors, (e.g. ketoconazole, itraconazole, voriconazole, posaconazole, fluvoxamine, nefazodone, nelfinavir, ritonavir) and/or strong CYP3A4 inducers (e.g. phenytoin, rifampin, rifabutin) within 14 days prior to randomization.
* History of another primary malignancy, with the exceptions of: non-melanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for >= 3 years
* Childs-Pugh A-C liver disease (Appendix II)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Uzzo, MD, Principal Investigator — PI
Locations (8):
- United States (8):
  - Yale School of Medicine, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering, New York, New York
  - Duke University Health System, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Geynisman DM, Kadow BT, Shuch BM, Boorjian SA, Matin SF, Rampersaud E, Milestone BN, Plimack ER, Zibelman MR, Kutikov A, Smaldone MC, Chen DY, Viterbo R, Joshi S, Greenberg RE, Malizzia L, McGowan T, Ross EA, Uzzo RG. Sporadic Angiomyolipomas Growth Kinetics While on Everolimus: Results of a Phase II Trial. J Urol. 2020 Sep;204(3):531-537. doi: 10.1097/JU.0000000000001065. Epub 2020 Apr 6. PMID 32250730

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Everolimus)
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Everolimus)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 68 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
BMI [Median (Full Range); unit: kg/m^2] | 29.4 [22.4 to 42.6]
AML volume [Median (Full Range); unit: cc] | 47.3 [9.8 to 217.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Tumor Volume Reduction Greater Than 25%
Description: Measuring the efficacy and tolerability of everolimus by measuring the number of patients with tumor volume reduction greater than 25% in sporadic AMLs as measured by DCE MRI
Time Frame: 12 months
Population: Some participants experienced adverse events and were withdrawn from the study, and therefore tumor volume reduction was not measured in these patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Everolimus)
Number analyzed (Participants) | 10
Participants | 5

2. Secondary Outcome: Safety and Tolerability of Everolimus in Patients With Sporadic AML
Description: Number of participants with treatment-related adverse events requiring dose reduction or study withdrawal as assessed by Common Toxicity Criteria for Adverse Effects (CTCAE v4.0)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Everolimus)
Number analyzed (Participants) | 20
Participants | 10

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment (Everolimus)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Everolimus) (N=20)
chest pain (Cardiac disorders) | 1
flank pain (Gastrointestinal disorders) | 1
dysuria (Renal and urinary disorders) | 1
pneumonitis (Infections and infestations) | 1
heart palpitations (Cardiac disorders) | 1 — Not due to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Everolimus) (N=20)
oral mucositis (Infections and infestations) | 14 (20)
Alanine aminotransferase increase (Renal and urinary disorders) | 10
anemia (Blood and lymphatic system disorders) | 9
Aspartate aminotransferase increase (Renal and urinary disorders) | 9
fatigue (General disorders) | 7
Hypercholesterolemia (Blood and lymphatic system disorders) | 7
Maculopapular rash (Skin and subcutaneous tissue disorders) | 7
diarrhea (Gastrointestinal disorders) | 5
Leukocyte decrease (Blood and lymphatic system disorders) | 5
Hypertriglyceridemia (Blood and lymphatic system disorders) | 4
Pruritis (Skin and subcutaneous tissue disorders) | 4
constipation (Gastrointestinal disorders) | 3
Xerostomia (General disorders) | 3
Lymphocyte decrease (Blood and lymphatic system disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Metabolism + nutrional disorders - other (Metabolism and nutrition disorders) | 3
Dysgeusia (General disorders) | 3
cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Vascular disorders) | 3
Skin + subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 3
Chills (General disorders) | 2
fever (General disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 2
limb edema (Blood and lymphatic system disorders) | 2
UTI (Infections and infestations) | 2
Elevated creatinine (Renal and urinary disorders) | 2
Neutrophil decrease (Blood and lymphatic system disorders) | 2
headache (General disorders) | 2
Nervous system disorders - other (Nervous system disorders) | 2
pneumonitis (Infections and infestations) | 2
acneiform rash (Skin and subcutaneous tissue disorders) | 2
involuntary movements (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Lack of tissue to correlate response to molecular markers of aberrant mTOR pathways. Lack for serum everolimus levels. Clinical significance of 25% volume reduction unknown. Patient withdrawals and incomplete protocol imaging.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT02539459/Prot_SAP_000.pdf